CLINICAL TRIAL: NCT03337308
Title: A Randomized, Double-Blind, Parallel Group Study to Evaluate the Efficacy and Safety of Bempedoic Acid 180 Mg + Ezetimibe 10 Mg Fixed-Dose Combination Compared to Bempedoic Acid, Ezetimibe, and Placebo Alone in Patients Treated With Maximally Tolerated Statin Therapy
Brief Title: A Study Evaluating the Safety and Efficacy of Bempedoic Acid Plus Ezetimibe Fixed-Dose Combination Compared to Bempedoic Acid, Ezetimibe, and Placebo in Patients Treated With Maximally Tolerated Statin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002FDC-053
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Hyperlipidemias
Keywords: hyperlipidemia; heterozygous familial hypercholesterolemia; atherosclerotic cardiovascular disease; high cholesterol; ASCVD; HeFH; LDL
MeSH Terms: conditions — Hyperlipidemias; Atherosclerosis; Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BA 180 mg + EZE 10 mg FDC (Experimental): Bempedoic acid (BA) + ezetimibe (EZE) fixed-dose combination (FDC) 180 mg/10 mg tablets taken orally once daily for 12 weeks
  Interventions: Combination Product: Bempedoic Acid + Ezetimibe Fixed-Dose Combination; Drug: Placebos
- BA 180 mg (Experimental): Bempedoic acid (BA) 180 mg tablets taken orally once daily for 12 weeks
  Interventions: Drug: Bempedoic Acid; Drug: Placebos
- EZE 10 mg (Active Comparator): Ezetimibe (EZE) 10 mg overencapsulated tablets taken orally once daily for 12 weeks
  Interventions: Drug: Ezetimibe; Drug: Placebos
- Placebos (Placebo Comparator): Placebos to match identical bempedoic acid + ezetimibe fixed-dose combination (FDC) 180 mg/10 mg tablet, or identical bempedoic acid 180 mg tablet, or identical ezetimibe 10 mg capsule, taken orally, once daily for 12 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Combination Product: Bempedoic Acid + Ezetimibe Fixed-Dose Combination — bempedoic acid + ezetimibe FDC 180 mg/10 mg tablet
  Other Names: Bempedoic Acid + Zetia FDC; ETC-1002 + Zetia
  Arms: BA 180 mg + EZE 10 mg FDC
Drug: Bempedoic Acid — bempedoic acid 180 mg tablet
  Other Names: ETC-1002
  Arms: BA 180 mg
Drug: Ezetimibe — ezetimibe 10 mg overencapsulated tablet
  Other Names: Zetia
  Arms: EZE 10 mg
Drug: Placebos — placebo tablet or capsule to match bempedoic acid + ezetimibe fixed-dose combination (FDC) 180 mg/10 mg tablet, or bempedoic acid 180 mg tablet, or ezetimibe 10 mg capsule
  Other Names: Placebo

SUMMARY:
The purpose of this study is to determine if Bempedoic Acid (BA) + Ezetimibe (EZE) in a fixed-dose combination (FDC) is effective and safe versus its individual components and placebo in patients with elevated LDL cholesterol treated with maximally tolerated statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Require lipid-modifying therapy for primary or secondary prevention of cardiovascular disease
* Fasting LDL-C ≥ 130 mg/dL for primary prevention or LDL-C ≥ 100 mg/dL for secondary prevention (history of HeFH and/or ASCVD)
* Treated with maximally tolerated statin therapy at stable dose for at least 4 weeks prior to screening

Exclusion Criteria:

* Total Fasting Triglyceride ≥ 400 mg/dL
* Renal Dysfunction or nephrotic syndrome or history of nephritis
* Significant cardiovascular disease or cardiovascular event within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Haberman, MD, Study Director — Esperion Therapeutics, Inc.
Locations (5):
- United States (5):
  - PMG Research of McFarland, Ames, Iowa
  - Foundation Cardiology, Nashua, New Hampshire
  - PMG Research of Piedmont Healthcare, Statesville, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - PMG Research of Knoxville, Knoxville, Tennessee

REFERENCES:
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Background] Authors/Task Force Members:; Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WM, Vlachopoulos C, Wood DA, Zamorano JL. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias: The Task Force for the Management of Dyslipidaemias of the European Society of Cardiology (ESC) and European Atherosclerosis Society (EAS) Developed with the special contribution of the European Assocciation for Cardiovascular Prevention & Rehabilitation (EACPR). Atherosclerosis. 2016 Oct;253:281-344. doi: 10.1016/j.atherosclerosis.2016.08.018. Epub 2016 Sep 1. No abstract available. PMID 27594540
- [Background] Silverman MG, Ference BA, Im K, Wiviott SD, Giugliano RP, Grundy SM, Braunwald E, Sabatine MS. Association Between Lowering LDL-C and Cardiovascular Risk Reduction Among Different Therapeutic Interventions: A Systematic Review and Meta-analysis. JAMA. 2016 Sep 27;316(12):1289-97. doi: 10.1001/jama.2016.13985. PMID 27673306
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Derived] Ballantyne CM, Laufs U, Ray KK, Leiter LA, Bays HE, Goldberg AC, Stroes ES, MacDougall D, Zhao X, Catapano AL. Bempedoic acid plus ezetimibe fixed-dose combination in patients with hypercholesterolemia and high CVD risk treated with maximally tolerated statin therapy. Eur J Prev Cardiol. 2020 Apr;27(6):593-603. doi: 10.1177/2047487319864671. Epub 2019 Jul 29. PMID 31357887

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data are presented for the Full Analysis Set, comprised of all randomized participants. One participant was randomized but was not treated.
Groups:
- Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC: Participants received bempedoic acid + ezetimibe fixed-dose combination (FDC) 180 milligrams (mg)/10 mg tablets orally once daily for 12 weeks.
- Bempedoic Acid 180 mg: Participants received bempedoic acid 180 mg tablets taken orally once daily for 12 weeks.
- Ezetimibe 10 mg: Participants received ezetimibe 10 mg overencapsulated tablets orally once daily for 12 weeks.
- Placebo: Participants received placebo to match the bempedoic acid + ezetimibe fixed-dose combination (FDC) 180 mg/10 mg tablet, the bempedoic acid 180 mg tablet, or the ezetimibe 10 mg capsule, taken orally, once daily for 12 weeks.
Period: Overall Study
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
Started | 108 | 110 | 109 | 55
Completed | 103 | 103 | 104 | 53
Not Completed | 5 | 7 | 5 | 2
Not completed — Adverse Event | 2 | 3 | 3 | 1
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data are presented for the Full Analysis Set, comprised of all randomized participants. One participant was randomized but was not treated.
Groups:
- Placebo: Participants received placebo to match the bempedoic acid + ezetimibe FDC 180 mg/10 mg tablet, the bempedoic acid 180 mg tablet, or the ezetimibe 10 mg capsule, taken orally, once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo | Total
Number analyzed (Participants) | 108 | 110 | 109 | 55 | 382
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (9.97) | 65.2 (9.54) | 64.4 (8.91) | 65.6 (10.74) | 64.4 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 65 | 57 | 22 | 202
  Male | 50 | 45 | 52 | 33 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 33 | 32 | 20 | 117
  Not Hispanic or Latino | 76 | 77 | 77 | 35 | 265
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 20 | 19 | 16 | 7 | 62
  White | 85 | 90 | 91 | 48 | 314
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline was defined as the mean of the last 2 non-missing values from Week -2 (Screening Visit [Visit S1]) and predose Day 1/Week 0 (Treatment Visit 1 [Visit T1]). Population: After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all data from these sites removed.
  milligrams per deciliter (mg/dL)
    number analyzed (Participants) | 86 | 88 | 86 | 41 | 301
    (all) | 153.80 (40.526) | 145.13 (38.456) | 148.80 (41.839) | 152.80 (46.773) | 149.70 (41.162)
Non-high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the last 2 non-missing values from Week -2 (Screening Visit [Visit S1]) and predose Day 1/Week 0 (Treatment Visit 1 [Visit T1]). Population: After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all data from these sites removed.
  mg/dL
    number analyzed (Participants) | 86 | 88 | 86 | 41 | 301
    (all) | 188.22 (46.657) | 175.67 (40.474) | 180.18 (47.308) | 180.91 (49.720) | 181.26 (45.595)
Total cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the last 2 non-missing values from Week -2 (Screening Visit [Visit S1]) and predose Day 1/Week 0 (Treatment Visit 1 [Visit T1]). Population: After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all data from these sites removed.
  mg/dL
    number analyzed (Participants) | 86 | 88 | 86 | 41 | 301
    (all) | 237.32 (48.694) | 225.55 (43.165) | 231.41 (50.478) | 231.27 (50.210) | 231.36 (47.857)
Apolipoprotein B (apo B) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the predose Day 1/Week 0 (Visit T1) value. Population: After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all data from these sites removed. Only participants with available data were analyzed.
  mg/dL
    number analyzed (Participants) | 82 | 85 | 84 | 38 | 289
    (all) | 121.1 (30.85) | 113.4 (26.43) | 115.5 (31.30) | 115.1 (32.52) | 116.4 (29.98)
High-sensitivity C-reactive protein (hsCRP) [Median (Inter-Quartile Range); unit: milligrams per liter (mg/L)] — Baseline was defined as the predose Day 1/Week 0 (Visit T1) value. Population: After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all data from these sites removed. Only participants with available data were analyzed.
  milligrams per liter (mg/L)
    number analyzed (Participants) | 84 | 87 | 85 | 40 | 296
    (all) | 3.08 [1.68 to 6.20] | 2.91 [1.40 to 5.04] | 2.78 [1.30 to 5.89] | 3.01 [1.26 to 5.51] | 2.96 [1.40 to 5.78]
Triglycerides (TGs) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the last 2 non-missing values from Week -2 (Screening Visit [Visit S1]) and predose Day 1/Week 0 (Treatment Visit 1 [Visit T1]). Population: After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all data from these sites removed.
  mg/dL
    number analyzed (Participants) | 86 | 88 | 86 | 41 | 301
    (all) | 177.19 (94.904) | 156.65 (71.985) | 161.73 (79.924) | 144.59 (55.814) | 162.33 (79.973)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the last 2 non-missing values from Week -2 (Screening Visit [Visit S1]) and predose Day 1/Week 0 (Treatment Visit 1 [Visit T1]). Population: After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all data from these sites removed.
  mg/dL
    number analyzed (Participants) | 86 | 88 | 86 | 41 | 301
    (all) | 49.19 (14.566) | 49.89 (12.383) | 51.23 (15.902) | 50.40 (14.067) | 50.14 (14.256)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the mean of the LDL-C values from Week -2 and predose Day 1/Week 0. Percent change from baseline in LDL-C was analyzed using analysis of covariance (ANCOVA) with treatment group and randomization stratification as a factors and baseline LDL-C as a covariate. Percent change from baseline was calculated as: ([LDL-C value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100. For LDL-C, if measured LDL-C value was available, measured LDL-C was used.
Time Frame: Baseline; Week 12
Population: Full Analysis Set (FAS), also known as the intention-to-treat set, was defined as all randomized participants. After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all efficacy data from these sites removed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 86 | 88 | 86 | 41
Percent Change | -36.2 (2.56) | -17.2 (2.52) | -23.2 (2.18) | 1.8 (3.49)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Difference of Least Squares (LS) means = -38.0, 95% CI 2-sided [-46.5 to -29.6], Standard Error of Mean 4.32 — Standard Error of the Difference of Least Squares (LS) Means
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Bempedoic Acid 180 mg; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -19.0, 95% CI 2-sided [-26.1 to -11.9], Standard Error of Mean 3.60 — Standard Error of the Difference of LS Means
Statistical Analysis 3: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, ANCOVA; Difference of LS means = -13.1, 95% CI 2-sided [-19.7 to -6.5], Standard Error of Mean 3.37 — Standard Error of the Difference of LS Means

2. Secondary Outcome: Percent Change From Baseline to Week 12 in High-sensitivity C-reactive Protein (hsCRP)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for hsCRP. Baseline was defined as the predose Day 1/Week 0 value. Percent change from baseline in hsCRP was analyzed using a non-parametric analysis. Percent change from baseline was calculated as: ([hsCRP value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100.
Time Frame: Baseline; Week 12
Population: FAS. Only participants with available data were analyzed. After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice;therefore, analysis was completed with all efficacy data from these sites removed.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 80 | 81 | 79 | 39
Percent Change | -35.1 [-56.5 to -2.3] | -31.9 [-62.6 to 7.7] | -8.2 [-34.4 to 32.0] | 21.6 [-18.5 to 68.5]
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, Wilcoxon rank sum test — using alpha = 0.01; Location shift = -46.1, 99% CI 2-sided [-78.75 to -15.78], Standard Error of Mean 12.22 — Standard Error of the Hodges-Lehmann Median Difference
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p = 0.002, Wilcoxon rank sum test — using alpha = 0.02; Median Difference (Final Values) = -25.6, 98% CI 2-sided [-45.00 to -7.15], Standard Error of Mean 8.14 — Standard Error of the Hodges-Lehmann Median Difference
Statistical Analysis 3: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Bempedoic Acid 180 mg; Test type: Superiority; p = 0.734, Wilcoxon rank sum test — using alpha = 0.02; Median Difference (Final Values) = -2.6, 98% CI 2-sided [-21.35 to 16.25], Standard Error of Mean 8.08 — Standard Error of the Hodges-Lehmann Median Difference

3. Secondary Outcome: Percent Change From Baseline to Week 12 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for non-HDL-C. Baseline was defined as the mean of the non-HDL-C values from Week -2 and predose Day 1/Week 0. Percent change from baseline in non-HDL-C was analyzed using ANCOVA with treatment group and randomization stratification as a factors and baseline non-HDL-C as a covariate. Percent change from baseline was calculated as: ([non-HDL-C value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100.
Time Frame: Baseline; Week 12
Population: FAS. After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all efficacy data from these sites removed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 86 | 88 | 86 | 41
Percent change | -31.9 (2.23) | -14.1 (2.17) | -19.9 (2.05) | 1.8 (3.28)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority — using alpha = 0.01; p < 0.001, ANCOVA; Difference in LS mean = -33.7, 99% CI 2-sided [-43.9 to -23.4], Standard Error of Mean 3.97 — Standard Error of the Difference of LS Means
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Bempedoic Acid 180 mg; Test type: Superiority; p < 0.001, ANCOVA — using alpha = 0.02; Difference in LS means = -17.8, 98% CI 2-sided [-25.1 to -10.5], Standard Error of Mean 3.12 — Standard Error of the Difference of LS Means
Statistical Analysis 3: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, ANCOVA — using alpha = 0.02; Difference in LS means = -12.1, 98% CI 2-sided [-19.1 to -5.0], Standard Error of Mean 3.03 — Standard Error of the Difference of LS Means

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol (TC)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for TC. Baseline was defined as the mean of the TC values from Week -2 and predose Day 1/Week 0. Percent change from baseline in TC was analyzed using ANCOVA with treatment group and randomization stratification as a factors and baseline TC as a covariate. Percent change from baseline was calculated as: ([TC value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100.
Time Frame: Baseline; Week 12
Population: FAS. Only participants with available data were analyzed. After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all efficacy data from these sites removed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 86 | 88 | 86 | 41
Percent change | -26.4 (1.90) | -12.1 (1.83) | -16.0 (1.59) | 0.7 (2.46)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — using alpha = 0.01; Difference of LS means = -27.1, 99% CI 2-sided [-35.1 to -19.1], Standard Error of Mean 3.11 — Standard Error of the Difference of LS Means
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Bempedoic Acid 180 mg; Test type: Superiority; p < 0.001, ANCOVA — using alpha = 0.02; Difference of LS means = -14.2, 98% CI 2-sided [-20.4 to -8.1], Standard Error of Mean 2.64 — Standard Error of the Difference of LS Means
Statistical Analysis 3: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p < 0.001, ANCOVA — using alpha = 0.02; Difference of LS means = -10.4, 98% CI 2-sided [-16.1 to -4.6], Standard Error of Mean 2.48 — Standard Error of the Difference of LS Means

5. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B (Apo B)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for apo B. Baseline was defined as the predose Day 1/Week 0 value. Percent change from baseline in apo B was analyzed using ANCOVA with treatment group and randomization stratification as a factors and baseline apo B as a covariate. Percent change from baseline was calculated as: ([apo B value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100.
Time Frame: Baseline; Week 12
Population: FAS. After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all efficacy data from these sites removed. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 82 | 85 | 84 | 38
Percent change | -24.6 (2.38) | -11.8 (2.18) | -15.3 (1.97) | 5.5 (2.97)
Statistical Analysis 1: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Placebo; Test type: Superiority; p < 0.001, ANCOVA — using alpha = 0.01; Difference of LS means = -30.1, 99% CI 2-sided [-39.9 to -20.3], Standard Error of Mean 3.81 — Standard Error of the Difference of LS Means
Statistical Analysis 2: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Bempedoic Acid 180 mg; Test type: Superiority; p < 0.001, ANCOVA — using alpha = 0.02; Difference of LS means = -12.8, 98% CI 2-sided [-20.3 to -5.3], Standard Error of Mean 3.23 — Standard Error of the Difference of LS Means
Statistical Analysis 3: Comparison: Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC vs Ezetimibe 10 mg; Test type: Superiority; p = 0.003, ANCOVA — using alpha = 0.02; Difference of LS means = -9.3, 98% CI 2-sided [-16.5 to -2.1], Standard Error of Mean 3.09 — Standard Error of the Difference of LS Means

6. Secondary Outcome: Percent Change From Baseline to Week 12 in High-density Lipoprotein Cholesterol (HDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for HDL-C. Baseline was defined as the mean of the HDL-C values from Week -2 and predose Day 1/Week 0. Percent change from baseline was calculated as: ([HDL-C value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100.
Time Frame: Baseline; Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 83 | 82 | 80 | 40
Percent change | -5.59 (12.269) | -5.40 (14.688) | -2.11 (11.590) | -0.54 (12.799)

7. Secondary Outcome: Percent Change From Baseline to Week 12 in Triglycerides (TGs)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for TGs. Baseline was defined as the mean of the TGs values from Week -2 and predose Day 1/Week 0. Percent change from baseline was calculated as: ([TGs value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100.
Time Frame: Baseline; Week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
Number analyzed (Participants) | 83 | 82 | 80 | 40
Percent change | -7.90 (25.633) | 7.94 (42.312) | -2.46 (33.402) | 5.47 (31.992)

ADVERSE EVENTS:
Time Frame: Up to approximately 14 weeks
Description: Treatment-emergent adverse events (TEAEs) are defined as adverse events (AEs) that began or worsened after the first dose of investigational medicinal product (IMP). The analysis was performed using the Safety Analysis Set which consists of all randomized participants who received at least 1 dose of blinded IMP.
Arm/Group | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC | Bempedoic Acid 180 mg | Ezetimibe 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/110 | 0/109 | 0/55
Serious Adverse Events (participants affected / at risk) | 8/107 | 7/110 | 10/109 | 1/55
Other Adverse Events (participants affected / at risk) | 26/107 | 27/110 | 26/109 | 12/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC (N=107) | Bempedoic Acid 180 mg (N=110) | Ezetimibe 10 mg (N=109) | Placebo (N=55)
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Coronary vascular graft stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Renal artery occlusion (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid 180 mg + Ezetimibe 10 mg FDC (N=107) | Bempedoic Acid 180 mg (N=110) | Ezetimibe 10 mg (N=109) | Placebo (N=55)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 4 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 6 | 4 | 1
Urinary tract infection (Infections and infestations) | 8 | 3 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 1
Headache (Nervous system disorders) | 2 | 4 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 3 | 5 | 2 | 0

LIMITATIONS AND CAVEATS:
After a Root Cause Analysis, three sites were found not to have followed Good Clinical Practice; therefore, analysis was completed with all data from these sites removed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT03337308/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT03337308/SAP_001.pdf